CLINICAL TRIAL: NCT01252459
Title: Amino-acid PET Versus MRI Guided Re-irradiation in Patients With Recurrent Glioblastoma Multiforme - a Randomised Phase II Trial
Brief Title: Amino-acid PET Versus MRI Guided Re-irradiation in Patients With Recurrent Glioblastoma Multiforme
Acronym: GLIAA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: Clinical Trials Center Freiburg (Unknown); University of Freiburg (Other); AG-NUK-RT (Unknown)
Responsible Party: Prof. Dr. med. Anca-Ligia Grosu, Department of Radiation Oncology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG NUK/RT 2010-1
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Recurrent Glioma (Glioblastoma Multiforme)
Keywords: AA-PET; T1-Gd-MRI; re-irradiation; recurrent glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: AA-PET based target volume delineation (Experimental): Experimental intervention (Arm A): High-precision re-irradiation. Target volume delineation based on AA-PET.
  Interventions: Radiation: Radiation Therapy
- Arm B: T1Gd-MRI based target volume delineation (Active Comparator): Control intervention (Arm B): High-precision re-irradiation. Target volume delineation based on T1Gd-MRI.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Experimental intervention (Arm A): High-precision re-irradiation (stereotactic fractionated radiation therapy (SFRT) and/or image guided radiation therapy, (IGRT), total dose 39 Gy, 3 Gy/d, 5x/ week. Target volume delineation based on AA-PET: GTV = AA uptake on PET, clinical target volume (CTV) = GTV+3mm, PTV = CTV+2mm
  Arms: Arm A: AA-PET based target volume delineation
Radiation: Radiation Therapy — Control intervention (Arm B): High-precision re-irradiation (SFRT and/or IGRT), total dose 39 Gy, 3 Gy/d, 5x/ week. Target volume delineation based on T1Gd-MRI: GTV = contrast enhancement on T1Gd-MRI, CTV = GTV+3mm, PTV = CTV+2mm
  Arms: Arm B: T1Gd-MRI based target volume delineation

SUMMARY:
This study is designed to evaluate the impact of radiotherapy target volume delineation based on AA-PET compared to target volume delineation based on contrast enhanced T1 weighted MRI (T1Gd-MRI) on the clinical outcome of patients with recurrent glioblastoma (GBM) as well as concerning therapeutic safety of the respective strategy.

DETAILED DESCRIPTION:
The higher sensitivity and specificity of amino-acids (L-[methyl-11C]-methionine, MET and O-(2-(1)-Fluoroethyl)-L-tyrosine, FET) positron emission tomography (AA-PET) in the diagnosis of gliomas in comparison to computed tomography (CT) and magnetic resonance imaging (MRI) was demonstrated in many studies and is the rationale for using them in target volume delineation of these tumors. Several clinical trials have demonstrated the significant differences between AA-PET and standard MRI in gross tumor volume (GTV) delineation for treatment planning.

A small prospective study in patients with recurrent high grade gliomas treated with stereotactic fractionated radiotherapy (SFRT) showed a significant improvement in survival when AA-PET or single photon emission tomography (AA-SPECT) were integrated in target volume delineation, in comparison to patients treated using CT/MRI alone (Grosu et al. 2005).

However, there are no randomized studies demonstrating the impact of AA-PET based irradiation treatment on the clinical follow-up in comparison to a traditional MRI/CT based treatment.

The goal of this study is to evaluate the impact of radiotherapy target volume delineation based on AA-PET (new strategy) on the clinical outcome of patients with recurrent glioblastoma (GBM) compared to target volume delineation based on contrast enhanced T1 weighted MRI (T1Gd-MRI) (traditional, established strategy). Concerning therapeutic safety, the topography of recurrence outside the primary target volume as well as the localization of necrosis after the re-irradiation will be determined. All side effects will be assessed by CTCAE version 4.0 and the safety analyses will present the worst grade of acute and late side effect by treatment arm for the whole study period (treatment and follow up). Patients will be asked to complete a quality of life (QoL) questionnaire (as assessed by the E-ORTC QLQ-C15 PAL) in regular time intervals.

This will be the first phase II randomized study evaluating the impact of molecular imaging on outcome after radiotherapy in brain tumor patients.

Another goal of the technical part of this study is the development of a standardized physical-technical methodology for the integration of AA-PET and other imaging biomarkers in tumor volume delineation in radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Local recurrence of GBM (WHO grade IV) and either not eligible for tumor resection or with macroscopic residual tumor after resection of recurrent GBM
* Recurrent tumor visible on AA-PET and MRI-T1-Gd with the diameter measuring 1 cm to 6 cm by either technique
* Target volume definition possible according to both study arms
* Previous radiation therapy of the primary with a maximal total dose 60 Gy
* At least 9 months since the end of pre-irradiation and randomisation
* At most 2 prior chemotherapy regimes
* Start of radiation therapy possible within 2 weeks from AA-PET
* Karnofsky Performance Score (KPS) ≥ 70%
* Age ≥ 18 years
* Written informed consent (IC) obtained

Exclusion Criteria:

* - No histological confirmation of Glioma at initial diagnosis)
* Recent (≤ 4 weeks before IC) histological result showing no tumor recurrence
* No recurrent tumor detectable on last AA-PET or MRI-T1-Gd
* Technical impossibility to use existing AA-PET for RT-planning
* No prior radiation treatment to the primary tumor
* less than 9 months between the end of first radiation treatment and randomisation
* more than 2 previous chemotherapy regimes or previous treatment with Avastin or other molecular targeted therapies
* less than 2 weeks between application of chemotherapy and randomisation
* additional chemotherapy or molecular targeted therapy or further surgery planned before diagnosis of further tumor progression after study intervention
* pregnancy, nursing or patient not willing to prevent pregnancy during treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 6 months after randomization

SECONDARY OUTCOMES:
Overall survival | 1 year after randomisation
  Kaplan-Meier: Performed on the per protocol population - all patients who are eligible and have started their allocated treatment
Volumetrical assessment of GTV and PTV | Interim analysis
  Volumetrical assessment of delineated gross tumor volume (GTV) and planning target volume (PTV) based on AA-PET vs. delineated GTV/PTV based on T1-Gd-MRI.
Topography of recurrence | Follow up (end of radiotherapy, 6 and 12 weeks after radiotherapy, then every 3 months)
  local relationship between recurrence and AA-PEt and MRI-derived TV
Localisation of necrosis after re-irradiation | Follow up (end of radiotherapy, 6 and 12 weeks after radiotherapy, then every 3 months)
Rate of long-term survivors | Follow up
  Rate of long-term survivors = Survivors > 1 year after randomisation
Quality of Life (QoL) | During Radiotherapy and Follow Up
  QoL assessed by the EORTC QlQ-C 15 PAL questionnaire
Rate of side effects | During Radiotherapy and Follow Up
  Assessed according to CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Anca-Ligia Grosu, Prof. Dr. med., Study Chair — Department of Radiotherapy, University Hospital Freiburg; Wolfgang Weber, Prof. Dr. med., Study Chair — Department of Nuclear Medicine, University Hospital Freiburg; Ursula Nestle, PD Dr. med., Study Chair — Department of Radiotherapy, University Hospital Freiburg
Locations (1):
- Department of Radiotherapy, University Hospital Freiburg, Freiburg I. Br., Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Grosu AL, Weber WA. PET for radiation treatment planning of brain tumours. Radiother Oncol. 2010 Sep;96(3):325-7. doi: 10.1016/j.radonc.2010.08.001. Epub 2010 Aug 20. PMID 20728952
- [Background] Grosu AL, Weber WA, Franz M, Stark S, Piert M, Thamm R, Gumprecht H, Schwaiger M, Molls M, Nieder C. Reirradiation of recurrent high-grade gliomas using amino acid PET (SPECT)/CT/MRI image fusion to determine gross tumor volume for stereotactic fractionated radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):511-9. doi: 10.1016/j.ijrobp.2005.01.056. PMID 16168843
- [Background] Grosu AL, Weber WA, Riedel E, Jeremic B, Nieder C, Franz M, Gumprecht H, Jaeger R, Schwaiger M, Molls M. L-(methyl-11C) methionine positron emission tomography for target delineation in resected high-grade gliomas before radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):64-74. doi: 10.1016/j.ijrobp.2005.01.045. PMID 16111573
- [Background] Grosu AL, Piert M, Weber WA, Jeremic B, Picchio M, Schratzenstaller U, Zimmermann FB, Schwaiger M, Molls M. Positron emission tomography for radiation treatment planning. Strahlenther Onkol. 2005 Aug;181(8):483-99. doi: 10.1007/s00066-005-1422-7. PMID 16044216
- [Background] Grosu AL, Lachner R, Wiedenmann N, Stark S, Thamm R, Kneschaurek P, Schwaiger M, Molls M, Weber WA. Validation of a method for automatic image fusion (BrainLAB System) of CT data and 11C-methionine-PET data for stereotactic radiotherapy using a LINAC: first clinical experience. Int J Radiat Oncol Biol Phys. 2003 Aug 1;56(5):1450-63. doi: 10.1016/s0360-3016(03)00279-7. PMID 12873691
- [Background] Grosu AL, Feldmann H, Dick S, Dzewas B, Nieder C, Gumprecht H, Frank A, Schwaiger M, Molls M, Weber WA. Implications of IMT-SPECT for postoperative radiotherapy planning in patients with gliomas. Int J Radiat Oncol Biol Phys. 2002 Nov 1;54(3):842-54. doi: 10.1016/s0360-3016(02)02984-x. PMID 12377338
- [Background] Weber WA, Wester HJ, Grosu AL, Herz M, Dzewas B, Feldmann HJ, Molls M, Stocklin G, Schwaiger M. O-(2-[18F]fluoroethyl)-L-tyrosine and L-[methyl-11C]methionine uptake in brain tumours: initial results of a comparative study. Eur J Nucl Med. 2000 May;27(5):542-9. doi: 10.1007/s002590050541. PMID 10853810
- [Background] Grosu AL, Weber W, Feldmann HJ, Wuttke B, Bartenstein P, Gross MW, Lumenta C, Schwaiger M, Molls M. First experience with I-123-alpha-methyl-tyrosine spect in the 3-D radiation treatment planning of brain gliomas. Int J Radiat Oncol Biol Phys. 2000 May 1;47(2):517-26. doi: 10.1016/s0360-3016(00)00423-5. PMID 10802381
- [Derived] Grosu AL, Weber WA, Graf E, Mix M, Nestle U, Schimek-Jasch T, Wiehle R, Mader I, Wurtemberger U, Langen KJ, Niyazi M, Paulsen F, Konig L, Giordano FA, Spehl I, Bernhardt D, Schymalla MM, Pottgen C, Semrau S, Brunner T, Hultenschmidt B, Krause BJ, Ciernik IF, Beck J, Baumert BG, Meyer PT, Urbach H, Popp I; GLIAA Study Group. O-(2-[18F]fluoroethyl)-L-tyrosine-PET-guided versus contrast-enhanced T1-weighted MRI-guided re-irradiation in patients with recurrent glioblastoma (GLIAA/NOA-10 ARO2013-01): a multicentre, open-label, randomised trial. Lancet Oncol. 2025 Dec 19:S1470-2045(25)00642-4. doi: 10.1016/S1470-2045(25)00642-4. Online ahead of print. PMID 41429128
- [Derived] Oehlke O, Mix M, Graf E, Schimek-Jasch T, Nestle U, Gotz I, Schneider-Fuchs S, Weyerbrock A, Mader I, Baumert BG, Short SC, Meyer PT, Weber WA, Grosu AL. Amino-acid PET versus MRI guided re-irradiation in patients with recurrent glioblastoma multiforme (GLIAA) - protocol of a randomized phase II trial (NOA 10/ARO 2013-1). BMC Cancer. 2016 Oct 5;16(1):769. doi: 10.1186/s12885-016-2806-z. PMID 27716184